CLINICAL TRIAL: NCT03001037
Title: dorsaVi Back Pain and Movement Registry
Acronym: BPAM
Status: Suspended | Type: Observational
Why Stopped: Pending internal study review and potential protocol modification
Sponsor: dorsaVi Ltd (Industry)
Collaborators: International Spine, Pain and Performance Center (Other)
Responsible Party: Sponsor
Other Study IDs: 051626(27149)
Record Dates: First submitted 2016-12-19; First posted 2016-12-22 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain
Keywords: Functional Outcome Measures; Wearable Sensors; ViMove; Low Back Pain; Range of Movement; Muscle Activity
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A - Low Back Pain: Group A:
  * Subject provides written authorization and/or consent per institution and geographical requirements
  * Subjects in Group A with a predominant complaint of Low back pain, with a minimum daily average VAS ≥ 30/100
  * Subjects in Group A are intended to be assessed with ViMove based on standard of care
  * Subject is willing to participate in follow-ups at 3, 6, 12 months post initial assessment
  Observational study, no intervention
- Group B - Without Low Back Pain: * Subject is without current low back pain
  * Subject does not have a history of low back pain lasting longer than 3 months in the past 12 months
  * Subject is willing to follow up 3 months post initial assessment
  Observational study, no intervention

SUMMARY:
This study will compare patients with low back pain (LBP) to age and gender matched controls to determine if there are differences between the two groups related to: range of movement, secondary outcomes (level of disability, quality of life, evidence of depression, anxiety or stress), movement patterns and demographic characteristics. The first phase will include a baseline and 3 month follow-up assessment of the LBP patients and controls, including demographic characteristics, outcome measures, and a physical assessment. The second phase is an ongoing phase with continued interim assessments of LBP patients only, at 6 and 12 months.

DETAILED DESCRIPTION:
The first phase of the study will use a non-randomized two-group prospective longitudinal study design (Group A subjects with LBP, Group B subjects without LBP). The second phase of the study will use a single-group prospective longitudinal study design (Group A, subjects with low back pain). A timeline and step-by-step detail of the study procedures for these phases are also described in Appendix B.

Group A which will include subjects with LBP, members of the research team will screen and attempt to consecutively enroll all patients who undergo assessment for low back pain at two clinical locations (International Spine Pain & Performance Center, and Synergy Manual Physical Therapy). The enrollment and baseline visit can occur at the same time. During enrollment each subject will privately be briefed on the purpose and involvement in the study and be allowed to ask questions and opt out if not interested. Informed consent will be reviewed and signed and each subject will be given a copy of the consent form (15 minutes). Since collection of "baseline data" (outcome measures and ViMove Assessment) is already considered standard clinical practice for subjects with low back pain at these clinical settings, providing informed consent would allow the researchers to access this information for purposes of the registry. A summary of the information collected at baseline will include: patient demographics/medical history (age, gender, pain episode duration, BMI, employment, marital status, comorbidities, co-interventions, ICD-10 LBP diagnosis), outcome measures (LBP movement pattern classification, LBP Classifier Questionnaire, QVAS for back and leg, Oswestry Disability index, START-Keele, Fear Avoidance Behavior Questionnaire, EuroQol-5D, DASS-21, patient perception of movement contribution to pain) (20 minutes), and an assessment (ViMove standard assessment, 30 sec chair test, 40m walk test) (25 minutes). See Appendix C.

Group B which will include subjects without LBP, members of the research team will recruit volunteers within the DC metro area using flyers posted on campus at the George Washington University, local DC metro gymnasiums and recreational centers, word of mouth and email list serves associated with educational programs within The George Washington University School of Medicine and Health Sciences. Subjects will be screened by phone for the presence or history of low back pain as well as other exclusion criteria. If the subject agrees to move forward with participation they will be asked to come to The George Washington University Program in Physical Therapy located at 2000 Pennsylvania Ave Suite 2000, NW Washington DC 20006, or International Spine Pain & Performance Center or Synergy Manual Physical Therapy. Enrollment and baseline visits can occur at the same time. During enrollment each subject will privately be briefed on the purpose and involvement in the study and be allowed to ask questions and opt out if not interested. Informed consent will be reviewed and signed and each subject will be given a copy of the consent form (15 minutes). Baseline data will then be collected which will include: subject demographics/medical history (age, gender, BMI, employment, marital status, comorbidities, co-interventions) and QVAS for back and leg, EQ-5D, DASS-21 (10 minutes) and ViMove standard assessment, 30 sec chair test, and 40m walk test (25 minutes). See Appendix C.

ViMove Testing (Groups A & B): The ViMove system (dorsaVi, Australia) which will be used to assess movement patterns and lumbar muscle activity in both groups during the ViMove standard assessment, 30 sec chair test, 40m walk test, is an inertial measurement system comprised of two wireless motion sensors containing a triaxial accelerometer, a triaxial gyroscope and a magnetometer, two wireless surface electromyography (EMG) sensors, and a small wireless recording device (RFD) that can be worn by the subject. The manufacturer reports average differences of < 1 degree for single plane, through range movements when comparing matched measurements from the ViMove and a Fastrak opto-electronic device (Charry, Umer et al. 2011). The ViMove motion sensors collect data at approximately 20 Hz.

When ViMove testing is performed for both groups, 4 sensors will be adhered to the subject's skin using customised biocompatible adhesives. The placement of the sensors is determined through the use of templates which have been validated as part of the FDA 510K application. During testing, the sensors communicate data wirelessly to the RFD which is connected to a computer running dorsaVi (ViMove software). Customised algorithms convert data generated by the software to meaningful biomechanical information, including measures such as range of movement, peak angles, speed of movement and muscle activation.

Subjects in Group A will follow-up with their healthcare provider based on standard clinical care practices. Enrolled subjects in Group A will undergo follow up at 3 months, 6 months and 12 months (45 minutes each session); these follow up visits may or may not coincide with a regular clinical office visit with their healthcare provider. Subjects in Group B will follow up at 3 months only (35 minutes).

Follow up will include completing outcome measures and an assessment as collected at baseline as well as collection of patient status, events, and protocol deviations.

Subjects may exit from the research project under the following circumstances:

* Subject chooses to withdraw (e.g. consent withdrawal)
* At the end of their follow-up period
* Investigator deems withdrawal is necessary (e.g. medically justified, failure of patient to maintain adequate registry compliance)
* Subject death
* Subject is no longer available for follow-up

ELIGIBILITY:
Inclusion Criteria:

Group A:

* Subject provides written authorization and/or consent per institution and geographical requirements
* Subjects in Group A with a predominant complaint of Low back pain, with a minimum daily average VAS ≥ 30/100
* Subjects in Group A are intended to be assessed with ViMove based on standard of care - Subject is willing to participate in follow ups at 3, 6, 12 months post initial assessment

Group B:

* Subject is without current low back pain
* Subject does not have a history of low back pain lasting longer than 3 months in the past 12 months
* Subject is willing to follow up 3 months post initial assessment

Exclusion Criteria:

* Subject who is, or is expected to be inaccessible for follow-up
* Subject with exclusion criteria required by local law
* Subject in whom movement assessment is contraindicated.
* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results
* Body mass index ≥ 35 - In Group B only, subjects who had a history of low back pain in the past 12 months which lasted > 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A:
  • Subject present with a predominant complaint of Low Back Pain, with a minimum daily average VAS ≥ 30/100
  Group B:
  • Subject is without current low back pain
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in Range of Movement from baseline | Baseline, 3 months, 6 months, and 12 months
  Maximal range of low back movement in sagittal and coronal planes

SECONDARY OUTCOMES:
Change in Muscle Activity from baseline | Baseline, 3 months, 6 months, and 12 months
  Surface EMG measurement of erector spinae muscle activity at L3 vertebra level
Change in Pain from baseline | Baseline, 3 months, 6 months, and 12 months
  Pain Score out of 100 as measured on VAS scale
Change in Keele StarT Back Tool scores from baseline | Baseline, 3 months, 6 months, and 12 months
  Screening test for Classification of severity of low back pain
Change in Fear Avoidance Beliefs Questionnaire responses from baseline | Baseline, 3 months, 6 months, and 12 months
  Measurement of fear and avoidance of physical activity and work related to low back pain
Change in Low Back Pain Classifier score from baseline | Baseline, 3 months, 6 months, and 12 months
  Questionnaire to classify low back pain into movement sub-categories based on movement related painful activities.
Change in EuroQol-5D scores from baseline | Baseline, 3 months, 6 months, and 12 months
  Quality of life measurement tool
Change in Oswestry Disability Index scores from baseline | Baseline, 3 months, 6 months, and 12 months
  Measurement of disability related to low back pain
ViMove 40m Fast Paced Walk | Baseline, 3 months, 6 months, and 12 months
  Time taken to complete test
Vimove 30 sec Sit to Stand Test | Baseline, 3 months, 6 months, and 12 months
  Count of repetitions of movement

CONTACTS AND LOCATIONS:
Overall Officials: Mehul J Desai, MD, Principal Investigator — International Spine, Pain and Performance Center
Locations (3):
- United States (3):
  - The George Washington University, Washington DC, Maryland
  - International Spine, Pain and Performance Center, Washington DC, Maryland
  - Synergy Manual Physical Therapy LLC, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Desai MJ, Jonely H, Blackburn M, Wanasinghage S, Sheikh S, Taylor RS. The Back Pain and Movement (B-PAM) registry; a study protocol. BMC Musculoskelet Disord. 2019 May 24;20(1):249. doi: 10.1186/s12891-019-2625-x. PMID 31122221